CLINICAL TRIAL: NCT00774904
Title: Adiponectin is Positively Associated With Insulin Resistance in Subjects With Type 2 Diabetic Nephropathy and Effects by Angiotensin Type 1 Receptor Blocker Losartan
Brief Title: Adiponectin and Insulin Resistance in Diabetic Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xi'an Jiaotong University (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: hui min Jin, shanghai No 3 people's hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADPN
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2008-10

CONDITIONS: Diabetic Nephropathy
Keywords: Type 2 Diabetes; Diabetic Nephropathy; Glucose Metabolism; Angiotensin II Type 1 Receptor Blockers
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 2 | interventions — Losartan

INTERVENTIONS:
Drug: Losartan — Angiotensin II Type 1 Receptor Blockers

SUMMARY:
Plasma adiponectin concentration is inversely associated with renal function. There is little literature on adiponectin levels and regulation by antihypertensive medication with an angiotensin II-receptor blocker (ARB), especially in subjects with type 2 diabetes in different stage of chronic kidney disease (CKD).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic nephropathy
* CKD at stage 1~4

Exclusion Criteria:

* Type 1 diabetes or nondiabetic renal disease
* An elevated plasma K level.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-04; Primary Completion 2007-10 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
GFR, HbA1c and the adiponectin concentration | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai No.3 people's hospital, Shanghai, China

REFERENCES:
- [Derived] Pan Y, Qiao QY, Pan LH, Zhou DC, Hu C, Gu HF, Fu SK, Liu XL, Jin HM. Losartan reduces insulin resistance by inhibiting oxidative stress and enhancing insulin signaling transduction. Exp Clin Endocrinol Diabetes. 2015 Mar;123(3):170-7. doi: 10.1055/s-0034-1395658. Epub 2014 Dec 11. PMID 25502581